CLINICAL TRIAL: NCT01383330
Title: Phase 1 Study of Daewon-ES(A) & Daewon-ES(B) in Healthy Male Volunteers Under Fed Condition
Brief Title: A Clinical Trial to Evaluate Pharmacokinetics of Daewon DW-ES(A) 625mg/5ml, Daewon DW-ES(B) 625mg/5ml and Megace 800mg/20ml in Healthy Male Volunteers Under Fed Condition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: gyujeong, Noh / professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DW-ES 1101
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers
Keywords: megesterol
MeSH Terms: interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Megace (Experimental): 800mg
  Interventions: Drug: megace
- DW-ES(A) (Active Comparator): 625mg
  Interventions: Drug: DW-ES(A)
- DW-ES(B) (Active Comparator): 625mg
  Interventions: Drug: DW-ES(B)

INTERVENTIONS:
Drug: megace — 800mg
  Arms: Megace
Drug: DW-ES(A) — 625mg
  Arms: DW-ES(A)
Drug: DW-ES(B) — 625mg
  Arms: DW-ES(B)

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics of Daewon DW-ES(A) 625mg/5ml, Daewon DW-ES(B) 625mg/5ml and Megace 800mg/20ml in healthy male volunteers under fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 55 years at screening.
* No significant congenital/chronic disease. No symptoms in physical examination.
* Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.

History of known hypersensitivity to drugs including valsartan and pitavastatin.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-09 (Estimated)